CLINICAL TRIAL: NCT06453655
Title: The Effect of Nursing Process Using Standard Nursing Terminologies in Colonoscopy Preparation of Outpatients on Bowel Cleansing
Brief Title: The Effect of Nurse Process on Bowel Cleansing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Humeyra Zengin, RN,PhD, Director of Nursing Services, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HUNP170977
Record Dates: First submitted 2024-05-30; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Colorectal Cancer; Colonoscopy Preparation; Boston Bowel Preparation Scale; Nursing
Keywords: Nursing Process; Standard Nursing Terminologies; NANDA-I Diagnoses; Nursing Intervention; Nursing Outcome
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Nursing Process

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Experienced endoscopists, who were unaware of the instructions given to the subjects, performed the colonoscopies. The endoscopist who performed the procedure added the visual assessment score to the patient's colonoscopy report, regardless of their participation in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This group was interviewed face to face one week before the day of the procedure and the nursing process was started to be applied. In the 3-day period before the procedure, the nursing process was continued with daily telephone follow-up. In the first face-to-face interview, nursing diagnoses and nursing outcome scales appropriate to the needs of the individual were determined and NOCs baseline measurements were made. NICs selected according to the nursing process were applied for 7 days. The last measurement of NOCs was made on the day of the procedure. In addition, BBPS scores calculated by the endoscopist during the procedure were taken from the patient file and recorded in the data collection form
  Interventions: Behavioral: Nursing Process
- Control Group (No Intervention): This grup nursing diagnoses and expected nursing outcomes (NOC) appropriate to the needs of the individual were selected in a face-to-face interview 1 week before the procedure. The baseline measurements of NOCs were made. On the trading day, the after measurement of NOCs was made. But nursing process was not applied to this group.

INTERVENTIONS:
Behavioral: Nursing Process — In the first step of the nursing process, nursing diagnoses NANDA-I and nursing outcomes (NOC) appropriate to the needs of the individual were selected. Immediately afterwards, the baseline measurements of NOCs were made. In the second stage, nursing interventions were determined in line with the selected diagnoses and started to be implemented. Instructions for the implementation of the selected NICs were reminded by phone 3 days before the procedure appointment and compliance with colonoscopy preparation instructions was monitored. In the third stage, after measurement of the NOCs were performed on the day of the procedure. In addition, the BBPS scores calculated by the endoscopist during the procedure were taken from the patient file and recorded in the data collection form and the stages of the nursing process were completed.
  Arms: Intervention

SUMMARY:
Colonoscopy is still the gold standard method for the diagnosis and treatment of colon cancers. Preparation for colonoscopy is a complex processa (eg. restricted diet three days before the procedure and to drink large volumes of drog ) involving many steps. It has been shown that the symptoms experienced by patients during colonoscopy preparation have an impact on the quality of the colonoscopy procedure. Adequate bowel preparation is essential for successful colonoscopy imaging and to detect and remove existing polyps. aim of this study was to examine the effect of the nursing process applied by using standard nursing terminologies on colonoscopy preparation of outpatients on bowel cleansing.

This study was designed as a prospective, single-blind, randomized controlled trial. This study tested the hypothesis that the nursing process using thestandard nursing terminologies NANDA-I, NIC and NOC for colonoscopy preparation has an effect on adequate bowel cleansing.

DETAILED DESCRIPTION:
Nurses use standardized nursing language (SNL) to address complex relationships between presenting problems and individuals from a holistic perspective. The most widely used nursing diagnosis classification worldwide is NANDA-I, which includes nursing outcomes and interventions, respectively. In this study, after determining the nursing diagnosis specific to the colonoscopy procedure (NANDA-I), we evaluated which nursing outcomes (NOC) were appropriate for the patient's condition and then selected the nursing interventions (NIC) with the highest probability of achieving the desired outcome and implemented a nursing process. The study was conducted as a prospective, endoscopist-blinded, randomized controlled trial at a hospital-based outpatient endoscopy center. Eligible patients were randomized into two groups. Both groups received verbal and written instructions according to standard care, while the intervention group received a nursing process. After the interview, NANDA-I diagnoses were determined according to the needs of the individuals, and NOC scales appropriate to these diagnoses were selected and NOCs were first evaluated. According to the prepared nursing care plan, the nursing interventions selected in accordance with the diagnoses were reminded to the patients by phone and their compliance with the colonoscopy preparation instructions was monitored. When the patient came to the hospital for colonoscopy, face-to-face interviews were conducted, and final evaluations of NOC scales were performed. Primary outcomes included bowel preparation scores graded using the Boston Bowel Preparation Score (BBPS) and secondary outcomes included scores on NOCs selected according to the process of preparation for the colonoscopy procedure.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 to 70 years,
* Outpatients admitted to the Gastroenterology Department and Endoscopy Unit of Hacettepe University Adult Hospital
* First-time colonoscopy screening patients,
* Patients who agreed to participate in the study by signing informed consent one week before the appointment

Exclusion Criteria:

* They had suspected or diagnosed colorectal cancer
* Previous colon surgery,
* Emergency colonoscopy
* Pregnancy
* Breastfeeding
* Diagnosed mental illness
* Class 3-4 heart failure,
* Patients with hearing problems
* Chronic renal failure requiring dialysis
* A family member undergoing colonoscopy at the same time
* Muscle weakness due to cerebrovascular disease, or hemiplegia/plegia
* People who wanted to leave the study during the research
* Those who are simultaneously included in the working groups due to family affinity
* Those who cannot complete the colonoscopy procedure for various reasons

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2018-12-30 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Boston Bowel Preparation Scale (BBPS) score for adequacy of bowel cleansing in all segments (0-2 points for each segment), mean and percentage of total (0-9) scores | 3 days after the procedure
  The BBPS scale was used in this study to visually evaluate all parts of the bowel (right, transverse, and left colon). On this scale, 9 points indicate excellent cleaning, and 0 points indicate inadequate bowel cleaning. According to BBPS, bowel cleansing is adequate if the score value for each segment is ≥ 2 points and above and the total score for all segments is ≥ 6 points and above. BBPS score <6 indicates inadequate bowel preparation. This scale has been used in the center where the study was conducted, and endoscopists indicate the results of the scale in writing in the colonoscopy procedure reports.BBPS scores calculated by the endoscopist during the procedure were recorded in the digital patient file. After the digital reports were approved by the relevant physician within 3 days after the procedure, the BBPS score in the patient file was included in the data collection form

SECONDARY OUTCOMES:
NOC-1 Knowledge: Prescribed Diet (1802) | 7 days before and on the day of the colonoscopy procedure
  The level of understanding of information about the diet recommended by a health professional for a specific health condition (14 items were evaluated) Evaluated as frequency, condition and intensity by the Likert scale, being 1 the worst score and 5 best score
NOC-2 Knowledge: Medication (1808) | 7 days before and on the day of the colonoscopy procedure
  The level of understanding of the information conveyed about a particular treatment regimen (13 items were evaluated) Evaluated as frequency, condition and intensity by the Likert scale, being 1 the worst score and 5 best score.
NOC-3 Compliance Behavior-Prescribed Diet (1622) | 7 days before and on the day of the colonoscopy procedure
  Personal actions to follow the food and fluid intake recommended by a health professional for a specific health condition (11 items were evaluated) Evaluated as frequency, condition and intensity by the Likert scale, being 1 the worst score and 5 best score.
NOC-4 Compliance Behavior-Prescribed Medication (1623) | 7 days before and on the day of the colonoscopy procedure
  Personal actions to safely administer a medicinal product as recommended by healthcare professionals to take full advantage of the therapeutic effects specific to a particular condition (13 items were evaluated) Evaluated as frequency, condition and intensity by the Likert scale, being 1 the worst score and 5 best score.
NOC-5 Anxiety Level (1211) | 7 days before and on the day of the colonoscopy procedure
  Level of severity of anxiety, stress or uneasiness caused by an unidentified cause (13 items were evaluated) Evaluated as frequency, condition and intensity by the Likert scale, being 1 the worst score and 5 best score
NOC-6 Communication (0902) | 7 days before and on the day of the colonoscopy procedure
  Express, receive and interpret verbal, written and non-verbal messages (11 items were evaluated) Evaluated as frequency, condition and intensity by the Likert scale, being 1 the worst score and 5 best score.
NOC-7 Skin Integrity: Skin Mucous Membranes (1101) | 7 days before and on the day of the colonoscopy procedure
  Unpleasant sensory and emotional experience arising from actual or potential or described tissue injury, with sudden or slow onset of mild to severe intensity, constant or recurrent, without an anticipated or predictable termination (5 items were evaluated). Evaluated as frequency, condition and intensity by the Likert scale, being 1 the worst score and 5 best score.
NOC-8 Comfort Status Physical (2010) | 7 days before and on the day of the colonoscopy procedure
  Physical comfort with body sensations and homeostatic mechanisms (13 items were evaluated) Evaluated as frequency, condition and intensity by the Likert scale, being 1 the worst score and 5 best score.
NOC-9 Sleep (0004) | 7 days before and on the day of the colonoscopy procedure
  Returning to the natural periodic pattern of the body's regeneration ( 11 items were evaluated) Evaluated as frequency, condition and intensity by the Likert scale, being 1 the worst score and 5 best score.

CONTACTS AND LOCATIONS:
Overall Officials: Humeyra Zengin, RN, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe Uviversity, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Study Protocol — https://doi.org/10.1097/MEG.0b013e328333fca6